CLINICAL TRIAL: NCT02540395
Title: Prospective Donor-specific Cellular Alloresponse Assessment for Immunosuppression Minimization in de Novo Renal Transplantation
Brief Title: Prospective Donor Specific T Response Measurment for IS Minimization in de Novo Renal Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Petra Reinke (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Petra Reinke, representative of the sponsor, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CELLIMIN; 2014-001325-33 (EudraCT Number)
Record Dates: First submitted 2015-08-19; First posted 2015-09-04 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Disorder Related to Renal Transplantation; Effects of Immunosuppressant Therapy
Keywords: Kidney transplantation; Immunosuppression; IFN-γ
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid; Steroids; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A: Standard of care (Active Comparator): Standard of care immunosuppressive regimen based on TAC (Prograf) (achieving 4-8ng/ml trough levels), MMF (Cellcept, Myfortic, Myfenax)(1gr bid) and steroids (6-methyl prednisolone, Urbason, Methypred) (according to KDIGO guidelines).
  All patients in group A recieve the tripple-drug IS as suggested by guidelines. In case of rejection the patients are treated with high dosage of Methypred and/or Thymoglobuline
  Interventions: Drug: Tacrolimus (for Group A); Drug: Mycofenolate mofetil (MMF) (for Group A); Drug: 6-methyl prednisolone (Steroids) (for Group A)
- Group B: "Low" Immunosuppression regimen (Experimental): (based on TAC monotherapy (Prograf) to achieve 8-10 ng/ml trough levels during the first 4 weeks after transplantation and 6-8 ng/ml thereafter, MMF (Cellcept, Myfortic, Myfenax) (1g bid) during the first 7 days post-transplant and stopped thereafter) and steroids (6-methyl prednisolone; Urbason, Methypred) (tapering until discontinuation on month 2 post-transplant).
  In contrast to Group A the patients are treated with a two drug IS combination consisting of Prograf and Methypred. In case of rejection the patients are treated with hifg dosage of Methypred and/or Thymoglobuline.
  Interventions: Drug: Tacrolimus (for Group B); Drug: MMF (mycophenolate mofetil) (for Group B); Drug: 6-methyl prednisolone (Steroids) (for Group B)

INTERVENTIONS:
Drug: Tacrolimus (for Group B) — Tacrolimus (for Group B) will be administered orally twice a day (bid). Tacrolimus (for Group B) will be initially given at the 0,1mg/kg bid to achieve a stable 12-hour trough level of 8-10 ng/mL during the first month after transplantation to progressively tapper to 6-8ng/ml thereafter.
  Other Names: Prograf
  Arms: Group B: "Low" Immunosuppression regimen
Drug: MMF (mycophenolate mofetil) (for Group B) — MMF (mycophenolate mofetil) will be administered orally to patients in group B at conventional doses (1gr/12h) before transplant procedure and during the first 7 days after transplant. For subjects who develop nausea, diarrhea, or other MMF(mycophenolate mofetil) -related gastrointestinal adverse effects (eg, symptoms fully assessed and deemed not to have an etiology other than intolerability to MMF), the MMF(mycophenolate mofetil) dose may be decreased to the maximally tolerated dose.
  Subjects unable to tolerate the reduced dose may be converted to mycophenolate sodium (Myfortic™) or to Myfenax.
  From day 8 on, patients will not receive MMF.
  Other Names: Cellcept; Myfortic; Myfenax
  Arms: Group B: "Low" Immunosuppression regimen
Drug: 6-methyl prednisolone (Steroids) (for Group B) — At the time of surgery, all patients will receive 500mg of 6-methyl prednisolone (Steroids, Urbason, Methypred).
  Patients in group B will receive 250mg of 6-methyl prednisolone (or equivalent) on day 2, 125 mg on day 3, 60 mg on day 4 and 30 mg on day 5. From day 6 on, patients will receive 0.25 mg/kg/d of 6-methyl-prednisolone (Steroids, Urbason, Methypred) until month 1, then tapering until discontinuation on month 2 will be performed.
  Other Names: Urbason; Methypred
  Arms: Group B: "Low" Immunosuppression regimen
Drug: Tacrolimus (for Group A) — The study group A will receive Tacrolimus (for Group A) (Prograf) to achieve 4-8 ng/ml trough levels during all the duration of the study.
  Tacrolimus (for Group A) (Tacrolimus) capsules should generally be administered on an empty stomach or at least 1 hour before or 2 to 3 hours after a meal, to achieve maximal absorption.
  Other Names: Prograf
  Arms: Group A: Standard of care
Drug: Mycofenolate mofetil (MMF) (for Group A) — Mycophenolate mofetil (MMF) (Cellcept, Myfortic, Myfenax) (for Group A) will be administered orally to patients in group A at conventional doses (1gr/12h). For subjects who develop nausea, diarrhea, or other Mycophenolate mofetil (MMF) (for Group A) -related gastrointestinal adverse effects (eg, symptoms fully assessed and deemed not to have an etiology other than intolerability to Mycophenolate mofetil (MMF) (for Group A), the Mycophenolate mofetil (MMF) (for Group A) dose may be decreased to the maximally tolerated dose.
  Subjects unable to tolerate the reduced dose may be converted to mycophenolate sodium (Myfortic™).
  The first dose of Mycophenolate mofetil (MMF) (for Group A) should be administered before transplantation.
  Other Names: Cellcept; Myfortic; Myfenax
  Arms: Group A: Standard of care
Drug: 6-methyl prednisolone (Steroids) (for Group A) — At the time of surgery, all patients will receive 500 mg of 6-methyl prednisolone (steroids for Group A).
  Patients in arm A will receive 20 mg/day of 6-methyl prednisolone (steroids for Group A) (or the equivalent) during the first 2 weeks after transplantation, then tapering to 15 mg from week 3 to week 4 to finally be maintained at 5mg/day.
  Other Names: Urbason; Methypred
  Arms: Group A: Standard of care

SUMMARY:
The main objective of the study is to demonstrate the utility and safety of the IFN-γ (Interferon Gamma) ELISPOT (Enzyme-linked immunosorbent spot) marker for the stratification of kidney transplant recipients into low and high IS (Immunosuppression) regimens. The enrichment study will test non-inferiority of low IS regimen compared to high IS regimen, assuming 10% of BPAR at 6-months in the control group, and allowing a non-inferiority limit of maximum 10%.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, age ≥18 years.
2. Subject must be a recipient of a first renal transplant from a deceased or living donor.
3. Subject must have a current documented PRA (Panel of reactive antibodies) <20% and no detectable anti-class I and II HLA (human leukocyte Antigens) antibodies by solid phase assay (Luminex®).
4. Subject is willing to provide signed written informed consent.
5. Women of Childbearing Potential (WOCBP) must be using a highly effective method of contraception (Pearl-Index < 1) to avoid pregnancy throughout the study in such a manner that the risk of pregnancy is minimized. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal [defined as amenorrhea ≥ 12 consecutive months; or women on hormone replacement therapy (HRT) with documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL]. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG (Human chorionic gonadotropin)) within 72 hours prior to the start of clinical trial.

Exclusion Criteria:

1. Subjects undergoing renal transplant with a current documented PRA >20% and/or detectable anti-class I and II HLA antibodies by solid phase assay (Luminex®).
2. CDC (complement dependent cytotoxicity) positive cross match.
3. Subjects receiving an allograft from a donor older than 65 years with elevated creatinine levels and/or treated diabetes.
4. Cold ischemia time (CIT) higher than 24h.
5. Subjects with a prior solid organ transplant (SOT), including renal re-transplantation, or receiving a concurrent SOT.
6. Patients previously treated with daclizumab or basiliximab.
7. Subjects with underlying renal disease of:

   * Primary focal segmental glomerulosclerosis.
   * Type I or II membranoproliferative glomerulonephritis
   * Atypical Haemolytic uremic syndrome (HUS) / thrombotic thrombocytopenic purpura syndrome.
8. Subject with Hepatitis B chronic infection and/or active infection by Hepatitis C virus (positive PCR (polymerase chain reaction result) at the moment of transplant.
9. Subjects with known human immunodeficiency virus (HIV) infection.
10. Patients with active systemic infection that requires the continued use of antibiotics.
11. Patients with neoplasia except localized skin cancer receiving appropriate treatment.
12. Patients with severe anemia (hemoglobin < 6g/dl), leucopenia (WBC (White blood cells) <2500/mm3), thrombocytopenia (platelets <80.000/mm3).
13. Hemodynamically instable patients even if their hemoglobin level counts > 6 g/dl.
14. Patients with intestinal pathology or severe diarrhoea that can hinder absorption according to medical criteria.
15. Subjects with a known hypersensibility to any of the drugs used in this protocol.
16. Subjects who have used any investigational drug within 30 days prior to enrolment in this clinical trial.
17. WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period, women who are pregnant or breastfeeding or women with a positive pregnancy test on enrolment.
18. Subjects who are legally detained in an official institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
assessment of anti-donor T-cell alloresponses using the IFN-γ ELISPOT test | 6 months
  Patients with a positive anti-donor IFN-γ ELISPOT assay result (>25 spots/300.000 PBMC (peripheral blood mononuclear cells )) will be ruled out of the study and patients with negative anti-donor IFN-γ ELISPOT test (<25 spots/300.000 PBMC) will be randomized in 2 different groups (1:1).
  The main objective of the study is to demonstrate the utility and safety of the IFN-γ ELISPOT marker for the stratification of kidney transplant recipients into low and high IS regimens.

SECONDARY OUTCOMES:
Differences across Treatment arms in eGFR (estimated glomerular Filtration rate) (ml/min) | after 3, 6 and 12 months
Differences across Treatment arms in Biopsy proven acute rejection rate (BPAR rate) | after 6 and 12 months
Differences across Treatment arms in subclinical rejection rate using renal allograft biopsy | after 3 and 12 months
Differences across Treatment arms in Prevalence of death, and graft loss | after 6 and 12 months
Differences across Treatment arms in Prevalence of metabolic and cardiovascular co-morbidity (new onset diabetes mellitus (NODAT, dyslipidaemias, hypertension) | 12 months
Differences across Treatment arms in Prevalence of subjects that remain MMF and steroid-free | after 6 and 12 months
Differences across Treatment arms in Prevalence of Acute and chronic histologic lesions assessed by the Bannf'11 score in protocol biopsies | after 3 and 12 months
Differences across Treatment arms in Prevalence of patients that remain on Therapy | after 12 months
Differences across Treatment arms in Distribution of patients in distinct chronic kidney diseases (CKD) stages | after 12 months
Differences across Treatment arms in treatment cost (cost/benefit) | after 1,3,6,12 and 24 months
Differences across Treatment arms in development of a Panel reactive T (PRT)-cell response platform to evaluate general anti-HLA T-cell Responses using ELISPOT | at pre-transplantation, 3, 6 and 12 months after transplantation as well as at time of BPAR
Differences across Treatment arms in assessment of anti-donor and anti-HLA antibodies by Solid phase assays (Luminex®) and B-cell ELISPOT | at pre-transplantation, 3, 6 and 12 months after transplantation as well as at time of BPAR
Differences across Treatment arms in different viral load (CMV, EBV, BKV) | at months 1, 2, 3, 6 and 12 after transplantation
Differences across Treatment arms in study of virus-specific T-cell responses (ELISPOT) | at at pre-transplantation, 3, 6 and 12 after transplantation
Differences across Treatment arms in prevalence of transcriptional genes by RT-PCR in PBMC (peripheral blood mononuclear cells ) | at pre-transplantation and months 1, 3, 6 and 12 after transplantation as well as at time of BPAR
Differences across Treatment arms in flow cytometry assessment of peripheral blood mononuclear cells (PBMC) | at pre-transplantation and months 1, 3, 6 and 12 after transplantation as well as at time of BPAR
Differences across Treatment arms in Quantitative analyses of urinary IP-10 (Interferon Gamma induced Protein) | at 4 weeks and at 3, 6 and 12 month after transplantation as well as at time of BPAR
Differences across Treatment arms in Assessment of protocol biopsies | at month 3 and 12 after transplantation
Differences across Treatment arms in MicroRNA assessment in sera and urine | at pre-transplantation and months 1, 3, 6 and 12 after transplantation
Differences across Treatment arms in evaluation of FOXP3 (Forkhead box P3) methylation degree at the TSDR (Treg-specific demethylated Region) | at pre-transplantation and months 1, 3, 6 and 12 after transplantation as well as at time of rejection

CONTACTS AND LOCATIONS:
Overall Officials: Josep M. Grinyó, Prof. Dr., Principal Investigator — Renal Transplant Unit, Department Nephrology Bellvitge Universitari Hospital
Locations (8):
- Institut klinické a experimentální mediciny, Prague, Prague 4, Czechia
- Centre Hospitalier Universitaire de Nantes, Nantes, France
- Germany (3):
  - Department Nephrology and BCRT, Charité Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Regensburg, Regensburg
- Academisch Medisch Centrum bij de Universiteit van Amsterdam, Amsterdam, Netherlands
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain
- Guy's Hospital, Great Maze Pond, London, United Kingdom